CLINICAL TRIAL: NCT00005101
Title: Study of Low Bone Mass in Premenopausal or Perimenopausal Women
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Columbia University (Other)
Other Study IDs: NCRR-M01RR00645-2738; CPMC-IRB-8414; CPMC-GCRC-2738
Record Dates: First submitted 2000-04-06; First posted 2000-04-07 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Osteoporosis
Keywords: disease-related problem/condition; osteoporosis; rare disease
MeSH Terms: conditions — Osteoporosis; Rare Diseases

SUMMARY:
OBJECTIVES:

I. Determine the possible causes of bone loss in premenopausal or perimenopausal women.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients undergo physical examination and complete history with emphasis on risk factors for osteoporosis and screening for occult secondary causes of osteoporosis through blood serum and 24 hour urine collection.

Patients with more than 6 months since prior bone mineral density measurements or who did not receive measurements at participating center, undergo dual energy x-ray absorptiometry over 30 minutes for bone mineral density measurements.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Low bone mass (T score less than -2.0) with no secondary cause on routine exam
* Premenopausal

OR

* Perimenopausal

--Prior/Concurrent Therapy--

* Chemotherapy: No prior or concurrent chemotherapeutic agents
* Endocrine therapy: No prior or concurrent glucocorticoids or suppressive doses of thyroid hormone
* Other: No prior or concurrent anticonvulsants

--Patient Characteristics--

* Hematopoietic: No multiple myeloma
* Other: No hyperparathyroidism No thyrotoxicosis No anorexia nervosa No Paget's disease of bone No rheumatoid arthritis No Cushing's syndrome No malabsorption syndrome No type I diabetes mellitus

Ages: 16 Years to 54 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1998-02

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Shane, Study Chair — Columbia University
Locations (1):
- Columbia University College of Physicians and Surgeons, New York, New York, United States